CLINICAL TRIAL: NCT01263470
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multicenter Study to Determine the Efficacy and Safety of SYR-322 in Subjects With Type 2 Diabetes in Japan
Brief Title: Efficacy and Safety of Alogliptin in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322/CCT-001; U1111-1118-3752 (Registry Identifier: WHO)
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; voglibose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Alogliptin 6.25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 12.5 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 50 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Voglibose 0.2 mg TID (Active Comparator)
  Interventions: Drug: Voglibose

INTERVENTIONS:
Drug: Alogliptin — Alogliptin 6.25 mg, tablets, orally, once daily for up to 12 weeks
  Other Names: SYR-322
  Arms: Alogliptin 6.25 mg QD
Drug: Alogliptin — Alogliptin 12.5 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: SYR-322
  Arms: Alogliptin 12.5 mg QD
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: SYR-322
  Arms: Alogliptin 25 mg QD
Drug: Alogliptin — Alogliptin 50 mg, tablets, orally, once daily for up to 12 weeks
  Other Names: SYR-322
  Arms: Alogliptin 50 mg QD
Drug: Voglibose — Voglibose 0.2 mg, tablets, orally, three times daily for up to 12 weeks.
  Other Names: Voglib; BASEN®
  Arms: Voglibose 0.2 mg TID
Drug: Placebo — Placebo-matching tablets, orally, once or three times daily for up to 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the dose-response relationships of alogliptin, once daily (QD) to an α-glucosidase inhibitor, three times daily (TID), to determine the optimal clinical dose for type 2 diabetic patients.

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

To evaluate the long-term safety and efficacy of alogliptin, participants in the present study could enter a long-term extension study SYR-322/OCT-001 (NCT01263496) that was planned separately.

ELIGIBILITY:
Inclusion Criteria:

* A glycosylated hemoglobin (HbA1c) value of 6.5% or more and below 10.0% 4 weeks after the start of screening(Week -4).
* A HbA1c differences within 10.0%* (*rounded off to the first decimal point) at the start of screening (Week -8) and 4 weeks after the start of screening (Week -4) from the HbA1c value at the start of screening.
* Was receiving a specific diet therapy and an exercise therapy (if any) for the last 4 weeks or longer before the start of screening (Week -8).

Exclusion Criteria:

* Received any antidiabetic drug within the last 4 weeks before the start of screening (Week -8) or during screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Department of Medicine, Study Director — Kawasaki Medical School
Locations (1):
- Okayama, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 54 investigative sites in Japan from 17 January 2007 to 22 December 2007.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus with uncontrolled blood glucose despite diet and exercise therapies were enrolled in one of 6, once-daily (QD) or three-times daily (TID) treatment groups.
Groups:
- Alogliptin 6.25 mg QD: Alogliptin 6.25 mg, tablets, orally, once daily for up to 12 weeks.
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily for up to 12 weeks.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily for up to 12 weeks.
- Alogliptin 50 mg QD: Alogliptin 50 mg, tablets, orally, once daily for up to 12 weeks.
- Voglibose 0.2 mg TID: Voglibose 0.2 mg, tablets, orally, three times daily for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Started | 75 | 79 | 84 | 80 | 79 | 83
Completed | 73 | 74 | 80 | 77 | 76 | 78
Not Completed | 2 | 5 | 4 | 3 | 3 | 5
Not completed — Adverse Event | 2 | 2 | 1 | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Participant Unavailability | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study Drug Non-compliance | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID | Total
Number analyzed (Participants) | 75 | 79 | 84 | 80 | 79 | 83 | 480
Age, Customized [Number; unit: participants]
  ≤ 64 years | 48 | 58 | 56 | 52 | 54 | 51 | 319
  ≥ 65 years | 27 | 21 | 28 | 28 | 25 | 32 | 161
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 25 | 17 | 24 | 27 | 135
  Male | 56 | 56 | 59 | 63 | 55 | 56 | 345

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Analysis based on last observation carried forward, where the last postbaseline double-blind observed value is carried forward and used for all subsequent scheduled time points where data is missing. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
percentage of Glycosylated Hemoglobin | 0.06 (0.456) | -0.51 (0.677) | -0.70 (0.572) | -0.76 (0.547) | -0.82 (0.474) | -0.16 (0.730)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.570, 95% CI 2-sided [-0.755 to -0.386]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.762, 95% CI 2-sided [-0.925 to -0.598]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.826, 95% CI 2-sided [-0.987 to -0.665]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.887, 95% CI 2-sided [-1.035 to -0.739]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.351, 95% CI 2-sided [-0.570 to -0.132]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.542, 95% CI 2-sided [-0.743 to -0.342]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.607, 95% CI 2-sided [-0.808 to -0.406]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.667, 95% CI 2-sided [-0.859 to -0.475]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 2).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 2 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
percentage of Glycosylated Hemoglobin | 0.00 (0.187) | -0.16 (0.153) | -0.17 (0.194) | -0.16 (0.187) | -0.15 (0.180) | -0.10 (0.204)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.158, 95% CI 2-sided [-0.213 to -0.104]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.174, 95% CI 2-sided [-0.234 to -0.114]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.160, 95% CI 2-sided [-0.219 to -0.100]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.153, 95% CI 2-sided [-0.212 to -0.095]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.059, 95% CI 2-sided [-0.116 to -0.003]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.075, 95% CI 2-sided [-0.136 to -0.014]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.061, 95% CI 2-sided [-0.121 to 0.000]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.054, 95% CI 2-sided [-0.114 to 0.006]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
percentage of Glycosylated Hemoglobin | -0.01 (0.336) | -0.34 (0.243) | -0.38 (0.309) | -0.35 (0.281) | -0.40 (0.284) | -0.16 (0.395)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.326, 95% CI 2-sided [-0.419 to -0.233]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.369, 95% CI 2-sided [-0.470 to -0.268]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.340, 95% CI 2-sided [-0.438 to -0.241]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.387, 95% CI 2-sided [-0.485 to -0.288]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.178, 95% CI 2-sided [-0.280 to -0.076]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.221, 95% CI 2-sided [-0.329 to -0.112]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.192, 95% CI 2-sided [-0.299 to -0.085]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.239, 95% CI 2-sided [-0.346 to -0.131]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
percentage of Glycosylated Hemoglobin | 0.00 (0.473) | -0.50 (0.432) | -0.61 (0.481) | -0.66 (0.432) | -0.69 (0.382) | -0.17 (0.634)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.500, 95% CI 2-sided [-0.644 to -0.356]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.614, 95% CI 2-sided [-0.763 to -0.464]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.660, 95% CI 2-sided [-0.804 to -0.516]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.695, 95% CI 2-sided [-0.832 to -0.559]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.325, 95% CI 2-sided [-0.494 to -0.156]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.438, 95% CI 2-sided [-0.610 to -0.267]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.485, 95% CI 2-sided [-0.654 to -0.315]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.520, 95% CI 2-sided [-0.683 to -0.357]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
mg/dL | 1.8 (28.26) | -13.8 (19.31) | -15.9 (20.26) | -14.3 (22.13) | -21.7 (25.65) | -8.0 (24.34)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -15.60, 95% CI 2-sided [-23.27 to -7.93]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -17.69, 95% CI 2-sided [-25.34 to -10.05]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -16.08, 95% CI 2-sided [-24.14 to -8.02]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -23.47, 95% CI 2-sided [-32.06 to -14.89]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.82, 95% CI 2-sided [-12.66 to 1.02]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -7.92, 95% CI 2-sided [-14.76 to -1.08]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -6.30, 95% CI 2-sided [-13.53 to 0.93]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -13.69, 95% CI 2-sided [-21.45 to -5.94]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
mg/dL | 8.4 (30.74) | -16.0 (20.88) | -20.9 (19.78) | -19.0 (20.64) | -23.3 (23.40) | -7.2 (26.77)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -15.60, 95% CI 2-sided [-23.27 to -7.93]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -17.69, 95% CI 2-sided [-25.34 to -10.05]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -16.08, 95% CI 2-sided [-24.14 to -8.02]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -23.47, 95% CI 2-sided [-32.06 to -14.89]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.82, 95% CI 2-sided [-12.66 to 1.02]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -7.92, 95% CI 2-sided [-14.76 to -1.08]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -6.30, 95% CI 2-sided [-13.53 to 0.93]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -13.69, 95% CI 2-sided [-21.45 to -5.94]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
mg/dL | 5.7 (27.40) | -12.0 (27.77) | -18.5 (22.71) | -18.6 (20.58) | -22.6 (27.60) | -3.5 (28.45)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -17.73, 95% CI 2-sided [-26.52 to -8.94]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -24.22, 95% CI 2-sided [-32.07 to -16.37]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -24.34, 95% CI 2-sided [-32.03 to -16.65]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -28.28, 95% CI 2-sided [-37.04 to -19.52]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -8.55, 95% CI 2-sided [-17.28 to 0.18]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -15.04, 95% CI 2-sided [-22.90 to -7.18]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -15.16, 95% CI 2-sided [-22.90 to -7.42]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -19.10, 95% CI 2-sided [-27.80 to -10.40]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
mg/dL | 5.6 (25.26) | -9.3 (32.36) | -14.6 (23.80) | -17.5 (20.71) | -22.6 (24.24) | -3.0 (27.69)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -14.92, 95% CI 2-sided [-24.19 to -5.64]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -20.17, 95% CI 2-sided [-27.86 to -12.48]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -23.07, 95% CI 2-sided [-30.41 to -15.73]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -28.17, 95% CI 2-sided [-36.05 to -20.29]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -6.27, 95% CI 2-sided [-15.60 to 3.06]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -11.52, 95% CI 2-sided [-19.41 to -3.64]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -14.42, 95% CI 2-sided [-22.04 to -6.80]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -19.52, 95% CI 2-sided [-27.61 to -11.43]

9. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 2).
Description: The change between the value of fasting C-peptide collected at week 2 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
ng/mL | 0.04 (0.772) | -0.11 (0.731) | 0.17 (0.756) | 0.18 (0.776) | 0.04 (0.619) | -0.11 (0.830)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.145, 95% CI 2-sided [-0.384 to 0.094]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.134, 95% CI 2-sided [-0.106 to 0.374]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.144, 95% CI 2-sided [-0.103 to 0.390]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.218 to 0.227]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.241 to 0.245]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.281, 95% CI 2-sided [0.038 to 0.524]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.291, 95% CI 2-sided [0.041 to 0.540]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.151, 95% CI 2-sided [-0.077 to 0.380]

10. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 4).
Description: The change between the value of fasting C-peptide collected at week 4 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
ng/mL | 0.01 (0.624) | -0.04 (0.634) | 0.02 (0.636) | 0.16 (0.697) | 0.05 (0.554) | -0.16 (0.767)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.045, 95% CI 2-sided [-0.245 to 0.156]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.185 to 0.210]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.158, 95% CI 2-sided [-0.053 to 0.369]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.140 to 0.235]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.122, 95% CI 2-sided [-0.097 to 0.341]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.179, 95% CI 2-sided [-0.036 to 0.395]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.325, 95% CI 2-sided [0.097 to 0.553]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.215, 95% CI 2-sided [0.006 to 0.423]

11. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 8).
Description: The change between the value of fasting C-peptide collected at week 8 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
ng/mL | 0.17 (0.882) | 0.05 (1.144) | 0.07 (0.792) | 0.24 (0.646) | 0.05 (0.592) | -0.05 (0.804)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.117, 95% CI 2-sided [-0.444 to 0.209]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.100, 95% CI 2-sided [-0.362 to 0.162]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [-0.166 to 0.324]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.117, 95% CI 2-sided [-0.355 to 0.121]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [-0.203 to 0.408]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.120, 95% CI 2-sided [-0.124 to 0.364]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.299, 95% CI 2-sided [0.071 to 0.526]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [-0.118 to 0.322]

12. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 12).
Description: The change between the value of fasting C-peptide collected at week 12 or final visit and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 79 | 84 | 79 | 79 | 83
ng/mL | -0.00 (0.692) | 0.04 (0.967) | 0.17 (0.609) | 0.25 (0.591) | 0.18 (0.696) | -0.02 (0.888)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.230 to 0.308]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.175, 95% CI 2-sided [-0.029 to 0.379]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.248, 95% CI 2-sided [0.044 to 0.453]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.186, 95% CI 2-sided [-0.035 to 0.407]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.236 to 0.340]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.188, 95% CI 2-sided [-0.044 to 0.421]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.261, 95% CI 2-sided [0.026 to 0.496]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.199, 95% CI 2-sided [-0.049 to 0.448]

13. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value).
Description: The change between the value of blood glucose collected at week 12 or final visit and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 80 | 78 | 76 | 79
mg/dL | -4.2 (42.10) | -28.1 (49.50) | -27.6 (43.88) | -44.8 (36.04) | -47.0 (32.66) | -22.7 (40.58)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -23.85, 95% CI 2-sided [-38.75 to -8.94]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -23.38, 95% CI 2-sided [-37.14 to -9.61]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -40.60, 95% CI 2-sided [-53.18 to -28.02]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -42.75, 95% CI 2-sided [-54.93 to -30.58]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.36, 95% CI 2-sided [-19.70 to 8.98]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -4.89, 95% CI 2-sided [-18.13 to 8.35]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -22.11, 95% CI 2-sided [-34.22 to -10.01]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -24.27, 95% CI 2-sided [-35.98 to -12.55]

14. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing - Area Under the Curve at 2 Hours (AUC (0-2)).
Description: as for outcome 13
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg·hr/dL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 80 | 78 | 76 | 79
mg·hr/dL | 5.6 (62.45) | -52.7 (75.51) | -55.0 (63.73) | -73.1 (51.21) | -81.8 (53.69) | -50.0 (62.49)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -58.31, 95% CI 2-sided [-80.79 to -35.83]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -60.66, 95% CI 2-sided [-80.84 to -40.47]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -78.72, 95% CI 2-sided [-97.03 to -60.40]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -87.43, 95% CI 2-sided [-106.26 to -68.60]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-24.69 to 19.23]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.07, 95% CI 2-sided [-24.85 to 14.70]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -23.13, 95% CI 2-sided [-41.16 to -5.11]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -31.84, 95% CI 2-sided [-50.36 to -13.33]

15. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing - Area Under the Curve at 2 Hours (AUC(0-2)).
Description: The change between the value of insulin collected at week 12 or final visit and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μU·hr/mL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 69 | 71 | 78 | 70 | 72 | 68
μU·hr/mL | -3.60 (12.940) | -0.74 (19.745) | 1.86 (15.602) | 4.12 (14.057) | -1.04 (23.333) | -15.40 (20.416)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 2.859, 95% CI 2-sided [-2.736 to 8.455]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 5.456, 95% CI 2-sided [0.748 to 10.165]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 7.715, 95% CI 2-sided [3.181 to 12.248]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 2.557, 95% CI 2-sided [-3.763 to 8.877]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 14.660, 95% CI 2-sided [7.924 to 21.396]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 17.257, 95% CI 2-sided [11.353 to 23.160]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 19.515, 95% CI 2-sided [13.629 to 25.401]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 14.357, 95% CI 2-sided [7.013 to 21.701]

16. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2).
Description: The change between the value of C-peptide collected at week 12 or final visit and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 80 | 78 | 76 | 79
ng·hr/mL | 0.01 (1.628) | 0.54 (1.787) | 0.77 (1.804) | 1.01 (1.957) | 0.97 (1.642) | -0.39 (2.091)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.535, 95% CI 2-sided [-0.019 to 1.089]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.764, 95% CI 2-sided [0.214 to 1.315]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.999, 95% CI 2-sided [0.418 to 1.580]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.959, 95% CI 2-sided [0.430 to 1.489]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.934, 95% CI 2-sided [0.315 to 1.552]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.163, 95% CI 2-sided [0.551 to 1.774]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.398, 95% CI 2-sided [0.759 to 2.036]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.358, 95% CI 2-sided [0.760 to 1.956]

17. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)).
Description: The change between the value of glucagons collected at week 12 or final visit and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg·hr/mL
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 72 | 75 | 79 | 78 | 76 | 79
pg·hr/mL | -15.8 (36.91) | -11.5 (37.45) | -4.5 (38.54) | -12.6 (47.23) | -19.5 (40.47) | -16.3 (52.26)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 6.25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 4.25, 95% CI 2-sided [-7.87 to 16.38]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 11.26, 95% CI 2-sided [-0.90 to 23.42]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 3.19, 95% CI 2-sided [-10.56 to 16.95]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 50 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -3.66, 95% CI 2-sided [-16.27 to 8.94]
Statistical Analysis 5: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 4.75, 95% CI 2-sided [-9.79 to 19.29]
Statistical Analysis 6: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 11.76, 95% CI 2-sided [-2.67 to 26.19]
Statistical Analysis 7: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 3.69, 95% CI 2-sided [-12.02 to 19.40]
Statistical Analysis 8: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -3.17, 95% CI 2-sided [-18.04 to 11.71]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Serious Adverse Events (participants affected / at risk) | 1/75 | 2/79 | 2/84 | 1/80 | 2/79 | 2/83
Other Adverse Events (participants affected / at risk) | 20/75 | 17/79 | 23/84 | 27/80 | 23/79 | 38/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Alogliptin 6.25 mg QD (N=79) | Alogliptin 12.5 mg QD (N=84) | Alogliptin 25 mg QD (N=80) | Alogliptin 50 mg QD (N=79) | Voglibose 0.2 mg TID (N=83)
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Alogliptin 6.25 mg QD (N=79) | Alogliptin 12.5 mg QD (N=84) | Alogliptin 25 mg QD (N=80) | Alogliptin 50 mg QD (N=79) | Voglibose 0.2 mg TID (N=83)
Flatulence (Gastrointestinal disorders) | 2 | 2 | 4 | 1 | 1 | 8
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 3
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 5 | 5 | 7 | 10 | 8 | 4
Bronchitis (Infections and infestations) | 1 | 3 | 2 | 0 | 2 | 0
Headache (Nervous system disorders) | 4 | 2 | 0 | 5 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 2 | 1 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.